CLINICAL TRIAL: NCT04639089
Title: The Effect of Platelet Rich Pasma on Strenal Healing Post Median Strenotomy in Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Hamdy Singab (Other)
Responsible Party: Sponsor-Investigator, Dr. Hamdy Singab, Professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD166/2020
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Surgical Procedures
Keywords: Cardiac Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Patient data will be collected preoperatively and intraoperatively and these risk factors will be studied Patients will be distributed to two equal groups. Demographic data : Age - gender - weight - BMI-DM-hist. of radiotherapy exposure -BIMA
  Intraoperative :
  We will apply 10cm plasma contain 1 million platlets on the sternal edge of only one group of them before sternal closure.
  post-operative The patients will be followed till being discharged from hospital and after the first 3 months after surgery sternal stability and absence of dehiscence will be primary out come measure
  Secondary end point :
  Severe form of sternal deheiscence After 3months: stability of sternum will be assessed By CT chest with 3D bone reconstruction and the value of bone density as aconfirmatory test
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We will apply 10cm plasma contain 1 million platlets on the sternal edge before sternal closure (Experimental): We will apply 10cm plasma contain 1 million platlets on the sternal edge before sternal closure
  Interventions: Drug: platlet rich plasma on sternal healing post median sternotomy
- We will apply 10cm saline on the sternal edge before sternal closure (Placebo Comparator): We will apply 10cm saline on the sternal edge before sternal closure
  Interventions: Drug: platlet rich plasma on sternal healing post median sternotomy

INTERVENTIONS:
Drug: platlet rich plasma on sternal healing post median sternotomy — Patient data will be collected preoperatively and intraoperatively and these risk factors will be studied Patients will be distributed to two equal groups. Demographic data : Age - gender - weight - BMI-DM-hist. of radiotherapy exposure -BIMA
  Intraoperative :
  We will apply 10cm plasma contain 1 million platlets on the sternal edge of only one group of them before sternal closure.
  post-operative The patients will be followed till being discharged from hospital and after the first 3 months after surgery
  Other Names: PRP

SUMMARY:
Platelet-rich plasma (PRP) is an autologous concentration of human platelets in a small volume of plasma.

Because it is an autogenous preparation, PRP is inherently safe and therefore free from concerns over transmissible diseases such as HIV and hepatitis.

Its power of regeneration already proved by orthopedics and dentists in their trials to regenerate cartilages .We will use it to know its ability to enhance healing of sternum in vulnerable patients to sternal dehiscence after open heart surgery .

DETAILED DESCRIPTION:
1. INTRODUCTION Successful healing of the sternum after open heart surgery is a complicated phenomenon because of the natural body ability often fails to efficiently repaired of the sternum in patients after open cardiac surgery (Everts 2006). Recent evidence based data suggested new modalities to increase the quality and accerelate sternal healing in high risk patients after open heart surgery vulnerable for early sternal dehiscence (Liu 2002) . PRP considers as an attractive alternative option in that manner. Marx and associates demonstrated the positive influence of PRP on bone regeneration and healing since 1998 (Marx 1998 ) . Autologous PRP carries minimal risk of infectious diseases transmission, immunologic reactions, and rejection. PRP with concentrations 4 to 5 folds of the normal average platelet (1,100,000 platelets/μl ) proved to have a remarkable increase in bone mineral density and regeneration . the market for PRP grows from $45 million in 2009 to more than $120 million by 2016 (Dawood 2018 ). Multiple factors affect the PRP efficacy in sternal bone healing and regeneration process. Platelet preparation before surgical application is an area of concern with PRP. For this issue, an appropriate anticoagulant must be used to prevent the early spontaneous activation of the platelets (Kassolis 2000 ). Several anticoagulants have been employed for PRP preparation including heparin, citrate, acid-citrate-dextrose solution A or anticoagulant citrate dextrose-A ,citrate-phos phate-dextrose ,citrate-theophylline-adenosine- dipyrimadole and ethylene diamine tetra- acetic acid moreover, several manual or automated systems have been designed for preparing PRP including clinical laboratory methods and kits (Carlson 2002). PRP produced by single- or double-step centrifugation technology via platelet-pheresis (autologous selective filtration )and the cell separators,However, these methods are rarely used nowadays, due to several factors including high cost, large volume of peripheral blood should be harvested from the patients, and potentially damage to the platelet (Dhurat 2014) . Commercially available PRP kits and devices differ in ease of use, one or two step centrifugation protocols, centrifugation speed, final PRP volume, platelet count and activation, platelet and growth factor concentrations, and final RBCs' and WBCs' count.Nevertheless, the cost of the commercial kits for PRP processing is still a challenge (Trebinjac 2020) .
2. AIM/ OBJECTIVES :

   To study the Effect of platlet rich plasma on sternal healing post median sternotomy in Patients undergoing open heart surgery
3. METHODOLOGY:

   * Type of Study: prospective clinical trial propensity matched comparative study
   * Study Setting: Patients refered to our Cardiothoracic department, Faculty of medicine, Ain Shams University and ain shams specialized hospital to perform open heart surgery who fulfill our inclusion charateria.
   * Study Period: It will be performed between march 2020 and january2022
   * Study Population:

     - Inclusion Criteria: Patients with one of which
     1. patients will under go open heart surgery with BMI >30 or
     2. diabetic patients
     3. patients with history of chest wall radiotherapy exposure or
     4. bilateral internal mammary artery harvesting .
     5. age > 70 years old -Exclusion Criteria:

     <!-- -->

     1. patient with history of open heart surgery
     2. patients with preoperative HB level <11
     3. All emergency and urgency cardiothoracic surgery
   * Sampling Method: prospective clinical trials propensity matched comparative study.
   * Sample Size: 50 patients
   * Ethical Considerations: All the patients will sign an informed consent for operation and for being involved in the research and follow up process .
   * Study Tools: platlets rich plasma
   * Preparation technique : ultra centrifuge technique
   * Study Procedures:

Patient data will be collected preoperatively and intraoperatively and these risk factors will be studied Patients will be distributed to two equal groups. Demographic data : Age - gender - weight - BMI-DM-hist. of radiotherapy exposure -BIMA

Intraoperative :

We will apply 10cm plasma contain 1 million platlets on the sternal edge of only one group of them before sternal closure.

post-operative The patients will be followed till being discharged from hospital and after the first 3 months after surgery sternal stability and absence of dehiscence will be primary out come measure

Secondary end point :

Severe form of sternal deheiscence After 3months: stability of sternum will be assessed By CT chest with 3D bone reconstruction and the value of bone density as aconfirmatory test

* Statistical Analysis:using the arithmetic mean, standard deviation using hypothesis student's "t" tests for quantitative data analysis, while qualitative data (ordinal, categorical) will be analyzed using The chi-square test (x2) (Fisher's Exact Test). For all statistical comparisons, a P value of <0.05 will be considered significant and a P value of <0.01 will be considered highly significant.
* Statistical Package:Data will be statistically analyzed using statistical package of social science (SPSS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of which

  1. patients will under go open heart surgery with BMI >30 or
  2. diabetic patients
  3. patients with history of chest wall radiotherapy exposure or
  4. bilateral internal mammary artery harvesting .
  5. age > 70 years old

Exclusion Criteria:

* patient with history of open heart surgery 2- patients with preoperative HB level <11 3-All emergency and urgency cardiothoracic surgery

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
sternal stability and absence of dehiscence | after the first 3 months of surgery
  Radiographic strenal healing score information was collected from 50 patients during clinical follow-up determined by CT chest 3D axial slices analysis at five locations ( manubrium, top of aortic arch, main pulmonary artery , aortic root and aortopulmonary window) using 5 - points quantitative scale 0:minimal healing
  1. no signs of healing
  2. mild healing
  3. moderate healing
  4. complete healing

CONTACTS AND LOCATIONS:
Overall Officials: hamdy singab, PHD, Study Director — faculty of medicine,ain shams unversity
Locations (1):
- Hamdy Singab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planning to make IPD available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available after 3 YEARS and for 2 years.
Access Criteria: IPD sharing access criertia including clinical researcher cardiac surgeons postgraduate investigator
URL: http://www.ctaegypt.org

REFERENCES:
- [Result] Carlson NE, Roach RB Jr. Platelet-rich plasma: clinical applications in dentistry. J Am Dent Assoc. 2002 Oct;133(10):1383-6. doi: 10.14219/jada.archive.2002.0054. PMID 12403541
- [Result] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595
- [Result] Kassolis JD, Rosen PS, Reynolds MA. Alveolar ridge and sinus augmentation utilizing platelet-rich plasma in combination with freeze-dried bone allograft: case series. J Periodontol. 2000 Oct;71(10):1654-61. doi: 10.1902/jop.2000.71.10.1654. PMID 11063400
- [Result] Liu Y, Kalen A, Risto O, Wahlstrom O. Fibroblast proliferation due to exposure to a platelet concentrate in vitro is pH dependent. Wound Repair Regen. 2002 Sep-Oct;10(5):336-40. doi: 10.1046/j.1524-475x.2002.10510.x. PMID 12406171
- [Result] Marx RE, Carlson ER, Eichstaedt RM, Schimmele SR, Strauss JE, Georgeff KR. Platelet-rich plasma: Growth factor enhancement for bone grafts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jun;85(6):638-46. doi: 10.1016/s1079-2104(98)90029-4. PMID 9638695
- [Result] Dawood AS, Salem HA. Current clinical applications of platelet-rich plasma in various gynecological disorders: An appraisal of theory and practice. Clin Exp Reprod Med. 2018 Jun;45(2):67-74. doi: 10.5653/cerm.2018.45.2.67. Epub 2018 Jun 29. PMID 29984206
- [Result] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694